CLINICAL TRIAL: NCT05919953
Title: Feasibility, Acceptability, and Usability of a Tele-rehabilitation Combining Immersive Virtual Reality Exercises and Therapeutic Education for Chronic Non-specific Neck Pain: A Mixed-methods Pilot Study.
Brief Title: Feasibility, Acceptability, and Usability of a Tele-rehabilitation Combining Immersive Virtual Reality Exercises and Therapeutic Education for Chronic Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VR NECK PAIN 2
Record Dates: First submitted 2023-05-04; First posted 2023-06-27 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Neck Pain
Keywords: Virtual reality; Therapeutic education; Tele-rehabilitation; Remote rehabilitation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality and therapeutic education (Experimental): Multimodal tele-rehabilitation consisting of therapeutic education and immersive virtual reality neck exercises.
  The duration of the intervention will be 6 weeks, including 5 virtual reality sessions (15-20 minutes per session, without supervision of the physiotherapist) and 1 teleconsultation session with a physiotherapist (30 minutes per session) per week.
  In addition, participants will receive several brochures to read on their own (therapeutic education). These brochures will be discussed with the physiotherapist during the teleconsultations.
  Interventions: Device: Virtual reality; Behavioral: Therapeutic education

INTERVENTIONS:
Device: Virtual reality — Immersive virtual reality neck exercises targeting relaxation, mobility, control, and speed of movement, using the Pico G2 4K headset.
Behavioral: Therapeutic education — Several brochures will be given to participants. These brochures will cover the general principles of pain, the persistence of pain, tips for managing chronic non-specific pain, and the use of immersive virtual reality in the rehabilitation of chronic non-specific neck pain.
  The information provided in the brochures will be discussed with the physiotherapist during the teleconsultations in order to individualize the therapeutic education.

SUMMARY:
Background: Several randomized controlled trials have already investigated the efficacy of virtual reality treatment for chronic neck pain, however no study to date has investigated multimodal tele-rehabilitation, combining both specific neck exercises in immersive virtual reality and therapeutic education, in subjects with chronic non-specific neck pain.

Objectives: The primary objective of this mixed-methods pilot study is to determine the feasibility, acceptability, and usability of tele-rehabilitation combining immersive virtual reality exercises and therapeutic education in people with chronic non-specific neck pain. Secondary objectives are: 1) to investigate changes in clinical outcomes (range of motion, pain intensity, neck disability, illness perceptions, kinesiophobia, impression of change) ; 2) to explore the subjects' experience of tele-rehabilitation.

Methods: The duration of the intervention will be 6 weeks, including 5 virtual reality sessions (15-20 minutes per session, without supervision of the physiotherapist) and 1 teleconsultation session with a physiotherapist (30 minutes per session) per week. Participants will be assessed quantitatively before and after the intervention, and qualitatively after the intervention.

Discussion: Study findings will provide evidence concerning the feasibility, acceptability, and usability of multimodal tele-rehabilitation for chronic non-specific neck pain, using immersive virtual reality. This study may strengthen the scientific evidence for the use of immersive virtual reality at home in the treatment of chronic non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years), men or women
* Chronic (> 3 months) non-specific neck pain (no specific cause responsible for the neck pain), with or without referred pain in the upper limbs or the head
* Neck Disability Index score greater than or equal to 5/50
* Numerical Pain Rating Scale score greater than or equal to 3/10 (average pain over the past week)
* To speak fluent French and to be able to provide informed consent

Exclusion Criteria:

* Age under 18 years
* Specific cause responsible for the neck pain (tumor/cancer, fracture, trauma, inflammatory disease, infection, compression or lesion of the spinal cord, surgery of the cervical spine, vascular pathology, neurological pathology, ligamentous lesion of the upper cervical spine, congenital disease of the cervical spine, chronic diffuse pain)
* Neck Disability Index score less than 5/50
* Numerical Pain Rating Scale score less than 3/10 (average pain over the past week)
* Signs of untreated sensorimotor dysfunction (vertigo, vestibular disorders/pathologies, etc.) that interfere with the use of virtual reality
* Visual problems (uncorrected myopia, limited vision after correction, eye surgery) that interfere with the use of virtual reality
* Altered comprehension, significant cognitive impairment, inability to speak French, deafness, pregnancy, inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention (retention rate) | At the end of the intervention (at 6 weeks)
  Retention rate (i.e., percentage of participants who completed the study).
Feasibility of the intervention (adhesion) | During the intervention (6 weeks)
  Adhesion to treatment (i.e., percentage of exercise sessions completed in relation to the total number of sessions prescribed, as well as the duration and frequency of the sessions).
Feasibility of the intervention (safety) | During the intervention (6 weeks)
  Safety (i.e., adverse events (type, frequency, severity) occurring during the intervention, assessed using a list of symptoms based on the Simulator Sickness Questionnaire and during the semi-structured interview).
Feasibility of the intervention (implementation at home) | At the end of the intervention (at 6 weeks)
  Implementation of the intervention at home (assessed during the semi-structured interview).
Feasibility of the intervention (online consultations) | At the end of the intervention (at 6 weeks)
  Number and duration of the online consultations.
Acceptability (satisfaction) of the tele-rehabilitation | At the end of the intervention (at 6 weeks)
  Satisfaction with the tele-rehabilitation (online consultations, weekly follow-up, virtual reality exercises,...) using 5-point Likert-scale questions (from "not at all satisfied" to "very satisfied") and during the semi-structured interview.
Usability of the virtual reality system and the online consultations | At the end of the intervention (at 6 weeks)
  Usability of the virtual reality system and the online consultations (assessed via the System Usability Scale (SUS) questionnaire and during the semi-structured interview). The SUS is a 10-item self-reported questionnaire assessing the usability of the interactive systems. Each item is scored from 1 ("do not agree at all") to 5 ("completely agree"). The total score ranges from 0 to 100, and higher scores reflect higher usability.

SECONDARY OUTCOMES:
Change in range of motion | Pre-intervention and at the end of the intervention (at 6 weeks)
  Cervical range of motion (CROM) will be assessed using the virtual reality headset.
Change in neck disability | Pre-intervention and at the end of the intervention (at 6 weeks)
  The Neck Disability Index (NDI) is a 10-item self-reported questionnaire assessing perceived neck disability by covering neck pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleep, and recreation. Each item is scored from 0 ("no disability") to 5 ("complete disability"). The total score ranges from 0 to 50, and higher scores reflect higher disability.
Change in pain intensity | Pre-intervention and at the end of the intervention (at 6 weeks)
  The Numeric Pain Rating Scale (NPRS) is a 11-point numeric horizontal scale assessing pain intensity from 0 ("no pain") to 10 ("worst possible pain"). NPRS will be used to measure the average pain intensity of the previous 7 days.
Change in kinesiophobia | Pre-intervention and at the end of the intervention (at 6 weeks)
  The Tampa Scale of Kinesiophobia (TSK) is a 17-item self-reported questionnaire used to assess kinesiophobia. Each item is scored from 1 ("strongly disagree") to 4 ("strongly agree"). The total score ranges from 17 to 68, and higher scores reflect increased kinesiophobia.
Change in illness perception | Pre-intervention and at the end of the intervention (at 6 weeks)
  The Brief Illness Perception Questionnaire (BIPQ) is a 9-item self-reported questionnaire assessing the cognitive and emotional representations of illness, illness comprehensibility, and the three most important causal factors in the patients illness (open-ended question). Each item (except the open-ended question) is scored from 0 to 10, where higher scores indicate stronger perceptions along that dimension. The total score ranges from 0 to 80, and higher scores reflect more negative perceptions.
Global perceived effect | At the end of the intervention (at 6 weeks)
  The Global Perceived Effect (GPE) will be assessed using a single 7-point Likert scale question about how the subject would describe him/herself in relation to before the intervention began (from 1 = "completely recovered" to 7 = "worse than ever").
Experiences of the intervention | At the end of the intervention (at 6 weeks)
  Experiences will be investigated during semi-structured interviews. These interviews will address the intervention (challenges, benefits, adhesion to treatment,...) and the virtual reality system (equipment, virtual environments, games,...).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pitance, PhD, Principal Investigator — Université Catholique de Louvain; Gaëtan Stoquart, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No